CLINICAL TRIAL: NCT03583268
Title: Determining the Appropriate Intensity of Vigorous Intensity Exercise to Prevent Post-exercise Hypoglycemia in Persons Living With Type 1 Diabetes
Brief Title: Determining the Appropriate Intensity of Exercise to Prevent Post-exercise Hypoglycemia in Persons Living With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B2014:095
Record Dates: First submitted 2015-03-18; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Physical activity; Hypoglycemia; Glucose variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moderate Intensity Exercise Alone (Active Comparator): 45 minutes of moderate intensity exercise at 45-55% of maximum aerobic capacity (active participants) or heart rate reserve (sedentary participants) used as a control condition. Participants will consume a glucerna bar at 10pm following this session.
  Interventions: Other: Exercise
- 70% Session (Experimental): 45 minutes of moderate intensity exercise interspersed with one minute bouts at 70% heart rate reserve every 4 minutes. Note: this session is not included for the active participants. Participants will consume a glucerna bar at 10pm following this session.
  Interventions: Other: Exercise
- 80% Session (Experimental): 45 minutes of moderate intensity exercise interspersed with one minute bouts at 80% of heart rate reserve every 4 minutes. Note: this session is not included for the active participants. Participants will consume a glucerna bar at 10pm following this session.
  Interventions: Other: Exercise
- 90% Session (Experimental): 45 minutes of moderate intensity exercise interspersed with one minute bouts at 90% of maximum aerobic capacity (active participants every two minutes) or heart rate reserve (sedentary participants every 4 minutes). Participants will consume a glucerna bar at 10pm following this session.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The intervention will be the different high intensity sessions. Time spent in hypoglycemia and glucose variability will be compared as follows: 70% vs. moderate, 80% vs. moderate, and 90% vs. moderate to see if high intensity is protective against hypoglycemia and provides lower glucose variability levels.

SUMMARY:
Over 300, 000 youth and young adults across Canada are living with Type 1 Diabetes (T1D) which is considered the most common endocrine condition. Physical activity offers numerous health benefits however the majority of persons living with T1D are physically inactive, primarily due to fear of low blood sugar (hypoglycemia). This fear of hypoglycemia continues to exist for physically active persons with T1D as no established physical activity guidelines exist. Several acute studies have used high intensity interval training as a way to reduce the risk of hypoglycemia as it has the ability to activate fight or flight hormones which can raise blood sugar; however the intensity needed to elicit this response is unknown.

The purpose of this project is to determine the acute effects of varying exercise intensities on the time spent in a low blood sugar range in 10 sedentary (VIGOR acute sedentary) and 16 physically active (VIGOR acute trained) individuals with T1D. Each participant will complete a maximal exercise test prior to the exercise sessions. Sedentary participants will complete 45 minutes of continuous moderate intensity exercise at 45-55% heart rate reserve (HRR) and three high intensity interval sessions with six one minute burst of high intensity at 70%, 80%, or 90% of HRR every four minutes. Active participants will complete 45 minutes of moderate intensity exercise at 45-55% of HRR and one high intensity interval session at 90% of HRR with intervals spaced every two minutes.

The investigators will track the blood sugar response to exercise using a device called a continuous glucose monitor (CGM) which records blood sugar every five minutes over a period of six days. The CGM will help determine which exercise intensity does a better job at reducing the time spent in a low blood sugar range. The information gained through this study will help individuals with T1D remain active without fear of low blood sugar and provide guidelines for professionals working with this population.

Adding high intensity bursts at 80% and 90% of maximum aerobic capacity (active participants) or heart rate reserve (sedentary participants) to a moderate intensity exercise session will significantly reduce the amount of time spent in a low blood sugar range in sedentary and active persons with T1D compared to moderate intensity exercise alone.

DETAILED DESCRIPTION:
Sedentary Arm: This portion of the study is complete. 10 participants completed the study in its entirety. Maximal exercise testing utilized a Parvomedics Metabolic cart to analyze oxygen consumption in ml/kg/min and maximum heart rate. Results from this test were used to estimate intensity using heart rate for the exercise sessions. Prior to each exercise session, participants arrived at 4:00 PM ate a Glucerna bar (to prevent drastic falls in glycemia with exercise) and had an IV inserted. A total of six blood samples were taken at each session at the following timepoints: (1) 0 mins-baseline, (2) 10 mins- end of warm up, (3) 35 mins-end of intervals, (4) 45 mins-end of exercise, (5) 75 mins-mid recovery, and (6) 105 mins-end of exercise. Each blood draw was sampled for glucose, cortisol, and growth hormone. Before exercise, blood glucose was measured on a handheld glucometer. If blood glucose was <5.7 mmol/L glucose was administered via Dex4 tablets. Exercise did not begin until blood glucose was at least 5.7 mmol/L. If blood glucose was greater than 16.7 mmol/L but less than 20.0 mmol/L ketones were tested on a urine ketone strip. If ketones were negative or trace exercise began.

The first exercise session was 45 minutes of moderate intensity exercise at 45-55% of heart rate reserve (HRR). The intensity determined from this session (speed and incline) was used as the recovery intensity for the high intensity sessions. The high intensity sessions were allocated in a random order from www.random.org where 1=70%, 2=80%, and 3=90%. Each high intensity session started with 10 minutes of moderate intensity exercise (at the same speed and incline from the first session) and six one minute bursts of high intensity every four minutes followed by a 10 minute cool down.

Because of the small sample size and non-normal glucose profiles, data was analyzed using a Friedman analysis of variance (non-parametric test).

Active Arm: This portion is still recruiting participants. The procedures for this experiment are very similar to the sedentary component. Blood glucose targets prior to exercise are the same however no blood samples will be taken. Participants will arrive at the lab for 4:30 PM and eat a Glucerna bar (to avoid drastic falls in glycemia with exercise). The two exercise sessions, moderate and 90%, will be allocated in a random order from a coin flip where heads is moderate exercise and tails is the 90% intervals. The moderate intensity session will consist of 45 minutes of exercise at 45-55% of HRR. The 90% session will consist of 15 minutes of moderate intensity at 45-55% of HRR followed by six one minute bursts of exercise at 90% of HRR every two minutes followed by a 10 minute cooldown.

Data will be analyzed using a general linear model and logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Persons with type 1 diabetes
* Hemoglobin A1c <9.9%
* Diabetes duration >/= 2 years
* Sedentary Participants: participate in <150 minutes of moderate to vigorous physical activity per week
* Active Participants: regular performance of vigorous physical activity >3 times/week for over one year. Display a maximal oxygen uptake that is at least 40.9 ml/kg/min for females, and 49.3 ml/kg/min for males.

Exclusion Criteria:

* HbA1c ≥9.9% as the lack of compliance with insulin suggests they may not be able to comply with the prescribed exercise requirements
* Have frequent and unpredictable hypoglycemia as they will be at a greater risk of serious hypoglycemic events
* Had a change in insulin management strategy, including adoption of a pump within two months of enrolment or switching back to multiple daily injections in the last two months, as they may be at risk for a hypoglycemic event due to the novel insulin management approach
* Have conditions that would render vigorous intensity activity contraindicated including: uncontrolled hypertension: BP >150 mm Hg systolic or >95 mm Hg diastolic in a sitting position; severe peripheral neuropathy; or history of cardiovascular disease
* Cognitive deficit resulting in an inability to provide informed consent
* Are currently taking beta-blockers as this would limit the ability to achieve target heart rates within the prescribed range
* Are currently being treated with medications (other than insulin) that alter glucose metabolism (i.e. atypical antipsychotics, corticosteroids)
* Are women who are pregnant, breastfeeding, or planning to get pregnant
* Have a job or profession that involves shift work (working during the night time, and being asleep during the daytime, as this alters glucose levels.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percent time spent </= 3.9 mmol/L as measured by continuous glucose monitor | 12 hours post exercise (6:00 PM to 6:00 AM)
  The time spent </= 3.9 mmol/L is measured through the continuous glucose monitor and is represented as a percentage.

SECONDARY OUTCOMES:
Mean absolute glucose change (MAG-mmol/L/h) as measured by continuous glucose monitor | 12 hours post exercise (6:00 PM to 6:00 AM)
  Glucose variability will be measured using a continuous glucose monitor assessed through mean absolute glucose change (MAG) which is a measure of inter-day variability (mmol/L/h)
Continuous overall net glycemic action (CONGA-mmol/L) as measured by continuous glucose monitor | 12 hours post exercise (6:00 PM to 6:00 AM)
  CONGA will be measured using a continuous glucose monitor assessed through overall net glycemic action (CONGA) which is a measure of intra-day variability (mmol/L).

OTHER OUTCOMES:
Cortisol | two hours post exercise
  Cortisol levels are assessed to see if these values are protective against hypoglycemia. Measured by competitive immunoassay with biotinylated polyclonal antibody against cortisol. Sedentary group only.
Growth hormone | two hours post exercise
  Growth hormone levels are assessed to see if these values are protective against hypoglycemia. As measured by immunosorbent assay. Sedentary group only.
Muscle mass as assessed by DEXA | Baseline appointment ~20 minutes
  For active individuals only. Muscle mass will be measured using a DEXA scanner

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McGavock, PhD, Principal Investigator — University of Manitoba; Children's Hospital Research Institute of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Facebook page for recruitment — https://www.facebook.com/profile.php?id=100005449635221